CLINICAL TRIAL: NCT00300625
Title: Validation of the San Francisco Syncope Rule
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Adrienne Birnbaum, Prof, Dept of Emergency Medicine, Albert Einstein College of Medicine
Other Study IDs: 04-05-109C
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Syncope; Near Syncope
Keywords: Syncope; Near syncope; San Francisco Syncope rule
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Application of the San Francisco Syncope Rule

SUMMARY:
This study was designed to validate the "San Francisco Syncope Rule". This set of rules was derived by Quinn et. al. to help guide the treatment of patients evaluated in the Emergency Department who had an episode of syncope (passed out) or near syncope (almost passed out). A rule that considers patients with an abnormal ECG, a complaint of shortness of breath, hematocrit less than 30%, systolic blood pressure less than 90 mm Hg, or a history of congestive heart failure was shown predict with a good degree of accuracy which patients would have an adverse event and require admission.

DETAILED DESCRIPTION:
This study was designed to validate the "San Francisco Syncope Rule". This set of rules was derived by Quinn et. al. to help guide the treatment of patients evaluated in the Emergency Department who had an episode of syncope or near syncope.

A rule that considers patients with an abnormal ECG, a complaint of shortness of breath, hematocrit less than 30%, systolic blood pressure less than 90 mm Hg, or a history of congestive heart failure was shown predict with a good degree of accuracy which patients would have an adverse event/serious outcome and require admission. Serious outcomes include the following: death,myocardial infarction, arrhythmia, pulmonary embolism, stroke, subarachnoid hemorrhage, significant hemorrhage, or any condition causing a return ED visit and hospitalization for a related event.

In Quinn's derivation trial, the sensitivity of the rule was 96%.

ELIGIBILITY:
Inclusion Criteria: Acute syncope or near syncope as a reason for the ED visit

Exclusion Criteria: Altered mental status, alcohol or illicit drug-related loss of consciousness, Definite seizure, Transient loss of consciousness caused by head trauma

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne J Birnbaum, MD, Principal Investigator — Albert Einstein College of Medicine; E J Gallagher, MD, Study Chair — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Quinn JV, Stiell IG, McDermott DA, Kohn MA, Wells GA. The San Francisco Syncope Rule vs physician judgment and decision making. Am J Emerg Med. 2005 Oct;23(6):782-6. doi: 10.1016/j.ajem.2004.11.009. PMID 16182988